CLINICAL TRIAL: NCT04332276
Title: A New Concept of Continuous Dopaminergic Stimulation by Cerebroventricular Administration of A-dopamine (dopamine Stored in Anaerobia) for Severe Motor Fluctuations in Parkinson's Disease?
Brief Title: Dopaminergic RestauratIon by IntraVEntriculaire Administration
Acronym: DIVE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: InBrain Pharma (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018_49; 2020-000155-12 (EudraCT Number)
Record Dates: First submitted 2020-03-25; First posted 2020-04-02 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2022-10

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; dopamine; L-dopa related motor complications; dyskinesia; symptomatic treatment; disease modifying effect
MeSH Terms: conditions — Parkinson Disease; Dyskinesias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cerebroventricular administration of A- dopamine (Experimental): Cerebroventricular administration of dopamine prepared and stored in anaerobia
  Interventions: Drug: A-dopamine
- Optimized oral dopaminergic treatment (Active Comparator): Optimized oral dopaminergic treatment with L-dopa (at least 5 doses a day) with dopaminergic agonist, monoamine B inhibitor and catechol-o-methyl inhibitor (if tolerated) (A-dopamine replaced by saline un the pump during optimized oral dopaminergic treatment)
  Interventions: Drug: optimized oral treatment

INTERVENTIONS:
Drug: A-dopamine — During the phase 1 (titration), it is planned to increase dopamine by maximum 0.25 mg per hour over the daytime period, which corresponds to a maximum increase of 4.5 mg per day (based on the 18 hours of the daytime period, since nocturnal needs are much less important).
  Then, depending on tolerance and efficacy, conservative titration will be continued for a target dose of 30-87 mg per day.
  During the phase 2 (efficacy), the treatment will be maintained at the minimum effective dose, planned between 30 and 87 mg per day, for 30 days.
  Arms: Cerebroventricular administration of A- dopamine
Drug: optimized oral treatment — The patient will received his usual dopaminergic treatment.
  Arms: Optimized oral dopaminergic treatment

SUMMARY:
Prospective monocentric randomized controlled open-label proof-of-concept study in cross-over of two 1-month periods and a long-term follow-up period not to exceed September 30, 2023, with 2 groups: Intracerebroventricular A-dopamine versus optimized oral medical treatment in parkinsonian patients at the stage of severe motor complications (fluctuations and dyskinesias) related to oral L-dopa.

In this study it will be expected to: 1) a higher benefit on motor symptoms 2) without tachyphylaxis, 3) a good ergonomic of the intra-abdominal pump refilled with A-dopamine every two weeks as compared with the numerous daily L-dopa doses and 4) a good safety profile of this classical neurosurgical procedure.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the second most frequent neurodegenerative disorder worldwide. The loss of dopamine through denervation in the striatum as a result of progressive neuronal degeneration in the substantia nigra pars compacta (SNpc), is the primary neurotransmitter marker of the disease. Since dopamine does not cross the digestive mucosa or the blood brain barrier, its lipophilic precursor L-dopa has been employed and remains the pivotal oral medication. However, after persistent use over several years, many pharmacokinetic drawbacks contribute to the occurrence of motor fluctuations and dyskinesia. Indeed L-dopa has a short half-life, limited and variable reabsorption through the digestive and blood brain barriers and potentially harmful peripheral distribution. Moreover, L-dopa requires the aromatic L-amino acid decarboxylase for the synthesis of dopamine, which declines in the striatum with disease progression. Intermittent oral doses of L-dopa induce discontinuous stimulation of striatal dopamine receptors that in turn contribute to dysfunctional dopaminergic pathways. Thus, continuous dopamine administration is considered more physiologically appropriate by preventing oscillations in neurotransmitter concentration.

It has been previously demonstrated that intracerebroventricular (i.c.v.) administered dopamine with an anti-oxidant adjuvant (sodium metabisulfite; SMBS) transiently improved motor handicap and increased dopamine in rat brains with unilateral neurotoxin 6-hydroxydopamine (6-OHDA)-induced damage as well as 1-methyl-4-phenyl-1,2,3,6-tetrahydropyridine (MPTP) intoxicated monkeys. The clinical feasibility of this administrative route has been supported by two PD patient case reports of dopamine infusion to the frontal ventricle, whereby a reduction in motor handicap was observed. Indeed, human case reports described a good tolerance to dopamine infusion over 1 year with a smooth control of motor symptoms. However, both preclinical and clinical reports also highlight two overriding problems that prevented further development; occurrence of tachyphylaxis and oxidation of dopamine causing enhanced dopamine metabolism and oxidative stress.

These prior challenges had been overcome by demonstrating that dopamine oxidation can be avoided by preparing, storing and administering dopamine in very low oxygen conditions (<0.01% of O2 = anaerobia = A-dopamine). In vitro, a positive effect of dopamine was observed on non-oncogenic dopaminergic neurons (LHUMES) survival. In vivo, A-dopamine restored motor function and induced a dose dependent increase of nigro-striatal dopaminergic neurons in mice after 7 days of MPTP intoxication that was not evident with either dopamine prepared aerobically (O-dopamine) or in the presence of a conservator (sodium metabisulfite, SMBS) or L-dopa. In the 6-OHDA rat model, continuous circadian i.c.v injection of A-dopamine over 30 days also improved motor activity without occurrence of tachyphylaxis. This safety profile was highly favorable, as A-dopamine did not induce dyskinesia or behavioral sensitization as observed with peripheral L-dopa treatment. In MPTP monkeys, A-dopamine improved the doparesponsive motor symptoms without inducing any dyskinesia or tachyphylaxis during 2 months. Indicative of a new therapeutic strategy for patients suffering from L-dopa related complications with dyskinesia, continuous i.c.v of A-dopamine had greater efficacy in mediating motor impairment over a large therapeutic index without inducing dyskinesia and tachyphylaxis.

In addition, greater advances in programmable pumps now minimize tachyphylaxis by allowing administration of a lower effective dopamine dose in accordance with the circadian cycle. Of note, PD patients from previous studies received O-dopamine and at the same dose throughout a 24 hours cycle. Prior experience obtained from the use of an apomorphine pump and duodopa® has identified the need to differentiate between diurnal and nocturnal minimum efficient dose in order to avoid worsening motor fluctuations.

Thus, continuous circadian i.c.v. administration of dopamine close to the striatum is feasible, efficient and safe in models of PD, supporting clinical development of this strategy to be revisited in PD patients with L-dopa related complications with dyskinesia.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease at the stage of L-dopa-induced severe motor and non-motor complications
* Men or women over 18 years old
* Parkinson's disease according to MDS criteria
* Severe motor complications including motor fluctuations with at least 2 hours of Off and 1 hour of dyskinesias uncontrolled by optimized oral drug therapy, i.e. with at least 5 doses of L-dopa and the addition or trial of a dopaminergic agonist (if tolerated) per os or by apomorphine pump
* The patient meets the criteria for a second-line invasive treatment such as deep brain stimulation (subthalamic or medial pallidum) or intrajejunal administration of levodopa gel (Duodopa®).
* Patients with a contraindication or who prefer this invasive therapeutic alternative to the other two existing and validated therapies (subthalamic stimulation or Duodopa®) because of its advantages: lower theoretical risk of intracerebroventricular delivery compared to subthalamic stimulation and better ergonomics than Duodopa®, but with the disadvantage of an as yet unproven benefit.
* Social security
* Able to provide free and informed consent to participate in research
* Patient willing to comply with all study procedures and duration
* Patient not planning to change lifestyle (nutritionally, physically or socially) during study participation

Exclusion Criteria:

* Over 75 years of age
* Subjects not receiving at least 5 doses per day of oral dopaminergic therapy
* Subject without a prior trial of an apomorphine pump (of lower risk); apomorphine pump treatment being a failure or a contraindication or refused by the patient
* Psychiatric history using the semi-structured psychiatric interview with DSM IV MINI: decompensated bipolar illness, psychotic state, current severe depression. Dysthymia and an isolated history of depression are not exclusion criteria.
* Patient with parkinsonian dementia (DSM IV and MDS criteria and MOCA score < or equal to 22)
* Isolated patient, defined as the absence of a caregiver present at least 3 hours/day in the patient's home.
* History of a fall in the last 6 months and/or a score >1 on items 2.12 (Walking and balance) and/or 3.12 (Postural stability) of the MDS-UPDRS scale
* Presence of another serious pathology threatening short- or medium-term vital prognosis, malnourished or cachectic patient.
* Hemostasis disorders
* Cardiac rhythm disorders and/or heart failure not controlled by treatment
* Uncontrolled blood pressure release
* Breastfeeding and pregnancy
* Women of childbearing age without effective contraception
* Contraindication to general anaesthesia
* Taking treatments containing guanethidine or related compounds or non-selective and selective monoamine oxidase A inhibitors (iproniazid, moclobemide, toloxatone)
* Neurosurgical contraindication (severe cerebral atrophy, brain tumor, infarction or other cerebral pathology, CSF flow disorder)
* Contraindication to abdominal placement of a subcutaneous pump and catheter that impairs healing and transcutaneous filling (e.g. major obesity, skin pathology, etc.).
* Contraindication to MRI (pacemaker, claustrophobia, etc.) and/or intolerance to gadolinium
* Active infectious pathology (including Covid-19)
* Immunologically deficient pathology likely to promote superinfection of equipment
* Patients under guardianship or trusteeship
* Patient already participating in another therapeutic trial using an investigational drug or in an exclusion period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
Percent Time Over Target | Month 1 through Month 2
  This is the amount of time that the BKS was over target and is a representation of "OFF" time in the period from 09:00-18:00 and is the proportion of time that a subject's BKS is greater than the target used in this study (BKS=26). The PTO does not include periods of immobility.
The number of hours with either perfect control or with a slight slowdown on the 7-day schedule | follow up visits every 6 months until the deadline of September 30, 2023
  Primary endpoint of the long-term follow-up phase . This will be compared to that obtained in phase 2 to demonstrate the maintenance of long-term efficacy control.

SECONDARY OUTCOMES:
bradykinesia score | At baseline and during the last day of each month of assessment ( an average 4 months)
  BKS calculated every two minutes throughout the period of wearing the logger. The median value of these BKS over the period from 09:00-18:00 for the full recording period is known as the median BKS and this correlates with the UPDRS III assessed at the time of doing the Kinetigraph Connected Actimeter (PKG®, Globalkinetics)
dyskinesia score | At baseline and during the last day of each month of assessment ( an average 4 months)
  DKS is calculated every two minutes throughout the period of that the logger is worn. The median value of these DKS over the period from 09:00-18:00 for the full recording period is known as the median DKS and this correlates with the modified Abnormal Involuntary Movement Score assessed at the time of donning the Kinetigraph Connected Actimeter (PKG®, Globalkinetics)
The Percent Time Immobile | At baseline and during the last day of each month of assessment ( an average 4 months)
  PTI over the period from 09:00-18:00. Immobility means that the logger, while being worn by the subject was entirely still for a two-minute period. This has been shown to correlate with the polysomnographic recordings of sleep.
The Fluctuation Dyskinesia Score | At baseline and during the last day of each month of assessment ( an average 4 months)
  FDS estimates the amount of variability in bradykinesia and dyskinesia as measured by the PKG over the course of the 6 days of recording. It provides a measure of the extent of fluctuations in bradykinesia and dyskinesia.
The Percent Time Tremor | At baseline and during the last day of each month of assessment ( an average 4 months)
  PTT is the proportion of time in the period from 09:00-18:00 that a subject spends with tremor. Tremor is likely to be present if PTT score >1%.
Unified Parkinson's Disease Rating Scale part III | At baseline and during the last day of each month of assessment ( an average 4 months); and follow up visits every 6 months until the deadline of September 30, 2023
  The Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III. MDS-UPDRS Part III measures motor examination. Part III consists of 33 scores based on 18 items, and each question is anchored with five response scale from 0(normal) to 4(severe).
Abnormal Involuntary Movement Score | At baseline and during the last day of each month of assessment ( an average 4 months); and follow up visits every 6 months until the deadline of September 30, 2023
  The AIMS rates 10 items of involuntary movement, each item ranging from 0 (no dyskinesia) to 4 (severe dyskinesia). Items assess facial, oral, extremity, and trunk movements, as well as self-awareness of abnormal movements.
Unified Dyskinesia Rating Scale | At baseline and during the last day of each month of assessment ( an average 4 months); and follow up visits every 6 months until the deadline of September 30, 2023
  The scale provides measurements for 'on-dyskinesias' and 'off-dyskinesias' and contains recommendations for descriptions of each type of involuntary movement
Montreal Cognitive Assessment | At baseline and during the last day of each month of assessment ( an average 4 months); and follow up visits every 6 months until the deadline of September 30, 2023
  Cognitive function was assessed by using MoCA score. Cognitive impairment was considered present when MoCA scores were <26 .
Neuropsychiatric Inventory | At baseline and during the last day of each month of assessment ( an average 4 months); and follow up visits every 6 months until the deadline of September 30, 2023
  otal NPI score is defined as the sum of the individual category scores. Higher scores on NPI indicate a more frequent and/or severe presence of neuropsychiatric behavioral changes. The following domains will be included in the subscore: Depression/Dysphoria, Anxiety, Apathy/Indifference, Irritability/Lability, Agitation/Aggression, and Disinhibition.
parkinson anxiety scale | At baseline and during the last day of each month of assessment ( an average 4 months); and follow up visits every 6 months until the deadline of September 30, 2023
  This scale is a 12-item observer or patient-rated scale with three subscales, for persistent and episodic anxiety, and avoidance behavior.
Lille apathy rating scale | At baseline and during the last day of each month of assessment ( an average 4 months); and follow up visits every 6 months until the deadline of September 30, 2023
  The Lille apathy rating scale is a measure of apathy through nine domains (each corresponding to a clinical manifestation of apathy: everyday productivity, interests, taking the initiative, novelty seeking, motivation - Voluntary actions, emotional responses, concern, social life & self-awareness) and 33 queries. The interview is structured, with a precise scoring mode for each reply (-2 to 2); when an item does not apply to the patient or the reply cannot be classified, it is scored "0" (for non-applicable and/or non-classifiable) The scale's overall score ranges from -36 to +36, with highest scores reflecting apathy severity. 4 factorial sub-scores (intellectual curiosity, emotion, action initiation and self-awareness) are calculated from sub-scale scores.
Parkinson's Disease Behavioral Assessment | At baseline and during the last day of each month of assessment ( an average 4 months); and follow up visits every 6 months until the deadline of September 30, 2023
  It rates 21 items that have 0 to 4 options : 0 = absent 1 = mild 2 = moderate 3 = marked 4 = severe
Global Impression of change | At baseline and during the last day of each month of assessment ( an average 4 months); and follow up visits every 6 months until the deadline of September 30, 2023
  The clinician Global Impression of change provides a brief, stand-alone assessment of the clinician's view of the patient's global functioning prior to and after initiating a study medication. It ranges from severely impaired to dramatically improved.
the Schwab and England scale | At baseline and during the last day of each month of assessment ( an average 4 months); and follow up visits every 6 months until the deadline of September 30, 2023
  The Schwab & England activities of daily living evaluates patients' autonomy through a percentage ranging from 0% (=Vegetative functions such as swallowing, bladder and bowel functions are not functioning. Bedridden.) to 100% ( = Completely independent. Able to do all chores without slowness, difficulty or impairment. Essentially normal).
Epworth Sleepiness Scale Questionnaire | At baseline and during the last day of each month of assessment ( an average 4 months); and follow up visits every 6 months until the deadline of September 30, 2023
  Epworth Sleepiness Scale Questionnaire. Outcome measure is between 0 and 24 with a score between 0-8 indicating normal Daytime sleepiness, a score between 9-14 indicating mild sleep deficiency and a score above 15 an excessive daytime sleepiness.
Parkinson's Disease Sleep Scale | At baseline and during the last day of each month of assessment ( an average 4 months); and follow up visits every 6 months until the deadline of September 30, 2023
  his scale allows to self-rate and quantify the level of sleep disruption being experienced. It rates 15 items that have 0 to 4 options, 4 is the worth option.
Parkinson's Disease Quality of Life Questionnaire (PDQ39) | At baseline and during the last day of each month of assessment ( an average 4 months); and follow up visits every 6 months until the deadline of September 30, 2023
  Parkinson's Disease Quality of Life Questionnaire (PDQ-39): the 39-Item Parkinson's Disease Questionnaire (PDQ-39) is a commonly used measure of self-appraisal in PD. It is a measure of health status and quality of life, by assessing difficulties in 8 dimensions of daily living: mobility (10 items), activities of daily living (6 items), emotional well-being (6 items), stigma (4 items), social support (3 items), cognition (4 items), communication (3 items) and bodily discomfort (3 items). The frequency of each event is determined by selecting one of 5 options: never (scored 0) / occasionally (scored 1) / sometimes (2) / often (3) / always (4). Each dimension total score range from 0 to 100, with lower scores reflecting better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Moreau, MD,PhD, Principal Investigator — University Hospital, Lille; David DEVOS, MD, PhD, Study Chair — University Hospital, Lille
Locations (1):
- Hopital Roger Salengro, CHU Lille, Lille, France

REFERENCES:
- [Derived] Moreau C, Odou P, Labreuche J, Demailly A, Touzet G, Reyns N, Gouges B, Duhamel A, Barthelemy C, Lannoy D, Carta N, Palas B, Vasseur M, Marchand F, Ollivier T, Leclercq C, Potey C, Ouk T, Baigne S, Dujardin K, Carton L, Rolland AS, Devedjian JC, Foutel V, Deplanque D, Fisichella M, Devos D. Intracerebroventricular anaerobic dopamine in Parkinson's disease with L-dopa-related complications: a phase 1/2 randomized-controlled trial. Nat Med. 2025 Mar;31(3):819-828. doi: 10.1038/s41591-024-03428-2. Epub 2025 Jan 7. PMID 39775041